CLINICAL TRIAL: NCT01660815
Title: PET Whole Body Biodistribution Using Florbetapir (18F)
Brief Title: A Study of Florbetapir (18F) in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-J02; I6E-AV-AVBA (Other: Eli Lilly Japan)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

ARMS (1):
- Healthy Volunteers (Experimental): Cognitively normal, healthy volunteers at least 45 years of age.
  Interventions: Drug: florbetapir (18F)

INTERVENTIONS:
Drug: florbetapir (18F) — IV injection, 370 MBq (10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; Florbetapir F 18

SUMMARY:
This study will determine how florbetapir (18F) (18F-AV-45) radioactivity is distributed throughout the body of Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Are Japanese cognitively normal healthy males or females at least 45 years of age;
2. Give informed consent; and
3. Are able to lie still on the imaging table for periods up to one hour.

Exclusion Criteria:

1. Have had radiation exposure (PET, SPECT or CT scans) for experimental purposes within the last year;
2. Are claustrophobic or otherwise unable to tolerate the imaging procedure;
3. Have medical conditions or surgical history that would confound evaluation of dosimetry (e.g., liver disease, colectomy etc.);
4. Have current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following:

   1. cardiac surgery or myocardial infarction within the last 6 months;
   2. unstable angina;
   3. coronary artery disease that required a change in medication within the last 3 months;
   4. decompensated congestive heart failure;
   5. significant cardiac arrhythmia or conduction disturbance, particularly those resulting in atrial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status;
   6. severe mitral or aortic valvular disease;
   7. uncontrolled high blood pressure;
   8. congenital heart disease;
   9. clinically significant abnormal result on ECG, including but not limited to QTc>450 msec; Before enrolling a patient with any evidence of the above conditions, the investigator must contact the sponsor;
5. Have current clinically significant medical comorbidities, as indicated by history, physical exam, or laboratory evaluations that might pose a potential safety risk, interfere with the absorption or metabolism of the study medication or limit interpretation of the trial results. These include but are not limited to clinically significant hepatic, renal, pulmonary, metabolic or endocrine disease, cancer;
6. Have a history of drug or alcohol abuse within the last year, or prior prolonged history of abuse;
7. Have a history of epilepsy or convulsions, except for febrile convulsions during childhood;
8. Have clinically significant infectious disease, including AIDS or HIV infection or previous positive test for hepatitis B, hepatitis C, HIV-1, or HIV-2;
9. Have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session;
10. Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Females of childbearing potential must not be pregnant (negative serum β-HCG at the time of screening) or breastfeeding at screening. Females must agree to avoid becoming pregnant, and must agree to refrain from sexual activity or to use reliable methods of contraception such as prescribed birth control or IUD for 24 hours following administration of florbetapir (18F);
11. Have a history of severe drug allergy or hypersensitivity;
12. Received an investigational medication within the last 30 days or who have participated in a clinical trial with any experimental medication in the last 30 days.

    Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication;
13. Have known hypersensitivity to alcohol; and
14. In the opinion of the investigator, are otherwise unsuitable for a study of this type.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Kobe, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Cognitively normal, healthy volunteers at least 45 years of age.
  florbetapir (18F) : IV injection, 370 MBq (10mCi), single dose
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  Japan | 7

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Radiation Dosimetry
Description: Radiation dose values (millisieverts/megabecquerel [mSv/MBq]) were calculated for target organs, including the adrenals, brain, breasts, gall bladder wall, heart wall, kidneys, lower large intestine wall, liver, lungs, muscle, ovaries, osteogenic cells, pancreas, red marrow, skin, small intestine, spleen, stomach wall, testes, thymus, thyroid, total body, upper large intestine wall, urinary bladder wall, and uterus.
Time Frame: 0-360 minutes
Population: Analysis population includes the 6 subjects who completed the study and had valid imaging data for quantitative analysis.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Groups:
- 50-kg Model: Radiation dose estimate using a 50-kg model.
- 70-kg Model: Radiation dose estimate using a 70-kg model.
Arm/Group | 50-kg Model | 70-kg Model
Number analyzed (Participants) | 6 | 6
mSv/MBq
  Adrenals | 0.0186 (0.000990) | 0.0132 (0.000685)
  Brain | 0.0179 (0.00234) | 0.0157 (0.00207)
  Breasts | 0.0108 (0.00123) | 0.00759 (0.000843)
  Gallbladder wall | 0.310 (0.192) | 0.268 (0.167)
  Heart wall | 0.0247 (0.00453) | 0.0171 (0.00316)
  Kidneys | 0.0237 (0.00393) | 0.0177 (0.00291)
  Lower large intestine wall | 0.0210 (0.00245) | 0.0161 (0.00178)
  Liver | 0.0456 (0.0249) | 0.0313 (0.0169)
  Lungs | 0.0127 (0.000885) | 0.00844 (0.000516)
  Muscle | 0.0136 (0.000989) | 0.00987 (0.000723)
  Osteogenic cells | 0.0493 (0.00575) | 0.0327 (0.00377)
  Ovaries | 0.0194 (0.000880) | 0.0139 (0.000727)
  Pancreas | 0.0205 (0.00188) | 0.0150 (0.00151)
  Red marrow | 0.0221 (0.00182) | 0.0155 (0.00118)
  Skin | 0.00993 (0.00113) | 0.00730 (0.000823)
  Small intestine | 0.0364 (0.00668) | 0.0269 (0.00506)
  Spleen | 0.0151 (0.00134) | 0.0105 (0.00105)
  Stomach wall | 0.0165 (0.000991) | 0.0120 (0.000689)
  Testes | 0.0128 (0.00118) | 0.00913 (0.000910)
  Thymus | 0.0133 (0.00176) | 0.00931 (0.00125)
  Thyroid | 0.0130 (0.00203) | 0.00922 (0.00143)
  Total body | 0.0161 (0.000468) | 0.0117 (0.000320)
  Upper large intestine wall | 0.0397 (0.00805) | 0.0299 (0.00611)
  Urinary bladder wall | 0.0578 (0.0364) | 0.0442 (0.0276)
  Uterus | 0.0199 (0.00157) | 0.0146 (0.00123)
  Effective dose | 0.0207 (0.00266) | 0.0149 (0.00198)

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less